CLINICAL TRIAL: NCT05680025
Title: Effect of a Physical Exercise Intervention Based on the Transtheoretical Model, on Blood Pressure in Patients With Hypertension, Insured by Mexican Institute of Social Security, in the State of Aguascalientes
Brief Title: Effect of a Physical Exercise Intervention Based on the Transtheoretical Model on Blood Pressure
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Ximena Duque López, Doctor of Science, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R-2021-101-054
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: Physical exercise; Transtheoretical Model; Lifestyle
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will be invited to attend two workshops, where they will be given and have explained a guide to physical activity and one for diet for patients with hypertension. In addition to pharmacological treatment, this is the information given as part of conventional treatment patients with hypertension receive from health care personnel.
- Physical exercise intervention (Experimental): Promoting physical exercise. The intervention group will have access to training videos through social networks and infographics.
  Interventions: Behavioral: Physical exercise intervention; Behavioral: Workshops

INTERVENTIONS:
Behavioral: Physical exercise intervention — The intervention group will have access to training videos through social networks (WhatsApp and YouTube) and infographics. The mobile phone of each of the participants will allow send dates of workshops, link for videos, messages reminding to perform exercise routines.
  The training plan will be designed so the participants will achieve being physically active at the end of 6 months of intervention. Training will be planned to gradually, through 3 levels, increase the duration and intensity of exercises; they will have an important component of aerobic exercises and others for muscular strength. Each level of training will last two months; at each level the participants will be given 4 specific trainings and will be asked to perform two per week at level 1 and 2; and at the 3 level, 3 trainings per week.
  The strategy for promoting physical exercise is based on the social cognitive theory, in which the bases of the transtheoretical model are found.
  Arms: Physical exercise intervention
Behavioral: Workshops — Six workshops to promote the performance of physical activity. The workshops will be held with groups of 15 participants. During them, the work will be to promote motivation to perform physical exercise, sharing information about the health benefits, benefits for control of the disease, together creating planning of measurable, realistic goals; reinforcing behavior when the desired advances are made, monitoring progress (using a monthly self-report of exercise performed). The participants will be motivated and congratulated each time for goals reached, self-sufficiency will be reinforced as well as greater evaluation of the advantages of performing exercise against the barriers or negative aspects perceived by the participants. These activities will be performed according to the level of exercise performed by the individuals (stage of change).
  Arms: Physical exercise intervention

SUMMARY:
Background: Hypertension is a public health problem; the World Health Organization (WHO) estimates that more than 1280 million people suffer it. The treatment of said condition is pharmacological and non-pharmacological. Physical activity is part of the treatment, but unfortunately few adults can be classified as physically active. There is evidence that performing physical exercise reduces systolic blood pressure by up to 5 mm Hg, which has associated with reduced heart disease by up to 9%, ictus up to 14% and all-cause mortality by 4%. Lifestyle changing interventions, among them promoting exercise marked by a theory of behavior change, have shown positive results. Objective: To evaluate the effect of an intervention promoting the performance of physical exercise, with specific recommendations, based on the Transtheoretical Model, on systolic blood pressure and on the amount of exercise performed (minutes/week) in patients with hypertension aged 40 to 70 years, users of primary care in the Mexican Institute for Social Security (IMSS) in Aguascalientes. Material and methods: Randomized clinical trial, in which 442 patients with hypertension will participate. The control group will receive conventional care and recommendations for physical exercise and diet. The intervention group, in addition, will attend 6 workshops, one a month, which will promote performing physical exercise, with access given to videos of physical exercise routines, designed to gradually increase the exercise performed. At the start and end of the study, blood pressure, anthropometric measurements will be taken, through a questionnaire asking about sociodemographic data, performance of physical exercise, psychosocial factors regarding physical exercise, diet and adherence to pharmacological treatment. The characteristics of the study population by group will be described, and changes between baseline and final measurements compared, intra and intergroup, in the systolic blood pressure and minutes/week of physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension.
* Patients from 40 to 70 years old.
* IMSS primary care users at UMF No. 1, in Aguascalientes.
* Patients who agree to participate in the study.

Exclusion Criteria:

* Patients with hypertension that have a medical contraindication for performing physical exercise, or whose health status suggests an individualized, supervised exercise plan (angina, arrhythmia, chronic kidney disease, lupus erythematosus).
* Patients who have some mental alteration that impedes answering the questionnaires or adequately following the established strategy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure | At baseline and at the end of the intervention (6 months)
  This will be obtained through the difference in means between final systolic pressure (at 6 months from the start of the study) less the baseline.
  Blood pressure will be determined after the participant's repose for 5 minutes, in a sitting position with the back supported against the chair, feet on the floor, the right arm at the height of the heart. The bracelet appropriate to the size of the arm will be used. Before measuring blood pressure by auscultation, the first number will be measured by palpitation. After these procedures and with an interval of 1 to 2 minutes, four measurements will be taken by the auscultator method, inflating the hose to 30 mm Hg above the figure in which pulse disappears and deflating at a rate of 2 mm Hg per second. The first noise of Korotkoff will be taken to define systolic pressure, and the disappearance of the Korotkoff noise marks diastolic pressure. The average of the last two takes will be used.

SECONDARY OUTCOMES:
Minutes of physical exercise per week | At baseline and at the end of the intervention (6 months)
  For the quantification of physical activity in minutes/week, the Physical Activity and Sedentary Behavior Questionnaire (Q-APCS) from the Canadian Society of the Physiology of Exercise and the Global Physical Activity Questionnaire will be used. The questionnaires will be applied at the start and finish of the study.
  The Q-APCS is comprised of 7 questions about the number of days/week in a typical week that moderate and vigorous physical activity are performed, and on the duration in minutes of these activities, also asking about the number of days per week performing strength and muscular resistance exercise, and on the hours/day being seated, in work or school and during free time, and on the frequency light activities are performed when seated in sedentary behavior for various hours. Global Physical Activity Questionnaire includes questions about minutes/week during which physical activity is carried out in leisure time.
  From this information, the minutes/week are calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ximena Duque, DS, Principal Investigator — Instituto Mexicano del Seguro Social; Segundo Moran, DM, Study Chair — Instituto Mexicano del Seguro Social; Laura Torres, Study Chair — Instituto del Saber Montfort
Locations (1):
- Unidad de Medicina Familiar No. 1, Aguascalientes, Mexico

IPD SHARING:
Plan to Share IPD: No